CLINICAL TRIAL: NCT07145307
Title: Evaluation of a Personalised Digital Treatment for Adolescents With Anxiety Disorders - A Feasibility Trial in Routine Care
Brief Title: Personalized Digital Treatment for Adolescent Anxiety: A Feasibility Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Alcohol and Drug Research Western Norway (KoRFor) (Unknown); Research Centre for Digital Mental Health Services (Forhelse) (Unknown)
Responsible Party: Principal Investigator, Pia Rygg Hauge, Principal Investigator, Helse Stavanger HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sidekick - A Feasibility Trial; Søknadsid 39864 (Other Grant/Funding Number: Helse Vests forskningsmidler 2025)
Record Dates: First submitted 2025-08-05; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorders
Keywords: anxiety disorders; digital interventions; digital cognitive behavioral therapy; digital ad-on; digital adjunct; adolescents; feasibility trial; exposure therapy; mobile app
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sidekick (Experimental): Use of the Sidekick app as an ad-on to regular outpatient treatment.
  Interventions: Device: Sidekick

INTERVENTIONS:
Device: Sidekick — An app for adolescents used to plan, complete and evaluate exposure exercises completed between sessions at a children and adolescent mental health clinic (BUP)
  Other Names: App-facilitated exposure therapy; Digital cognitive behavioral therapy; Digital adjunct; Digital ad-on

SUMMARY:
The goal of this feasibility study is to test whether a new blended digital intervention for adolescents with anxiety disorders is feasible and acceptable for use, and to help plan future larger scale studies. The main questions it aims to answer are:

* A: Can the investigators recruit appropriate participants?
* B: How appropriate are the data collection procedures and outcome measures?
* C: Are the study procedures and interventions suitable for and acceptable to the participants?
* D: Does the research team have the resources and ability to manage the study and intervention?
* E: Does the intervention show promise of being successful for adolescents with anxiety disorders?

Participants will:

* Receive outpatient anxiety treatment, typically every other week or weekly.
* Use the Sidekick app as a homework supplement to plan, carry out, and evaluate exposure exercises between treatment sessions.
* Complete questionnaires before, during, after, and three months after using the app.
* Some participants and therapists will be invited to take part in qualitative interviews following the intervention.

DETAILED DESCRIPTION:
1. Study goals and objectives

   This project will investigate the feasibility of an app-facilitated exposure therapy for adolescents with anxiety. The primary objective is to contribute to the development of an efficient and personalized digital treatment. To meet this objective, the project aims i) evaluate the feasibility of Sidekick, a personalized digital treatment tool for patients with anxiety disorders, and ii) evaluate the user experience of digitally assisted exposure therapy on patient-clinician dyads.

   1.1 Short-term and long-term goals

   In the short-term, this project will implement an open, explorative trial of Sidekick in specialized clinical practice. In the long-term, the project will report, communicate and implement findings in clinical and user settings. If results indicate that the blended intervention is feasible and acceptable, the next step is to seek funding and perform a large-scale, national randomized controlled trials (RCT) of a blended treatment protocol for anxiety in adolescents.
2. Feasibility

2.1 Study design, choice of methodology and analysis

To meet the goals of this project, the investigators will conduct a single-arm feasibility trial of the app Sidekick in a blended intervention for anxiety disorders in adolescents. The open trial will include data from patients and their clinicians. The study will provide feasibility insights, determining the practicality of implementing the tool within the outpatient clinic. It will highlight usability and acceptance, as well as preliminary effectiveness of the app. User and therapist feedback will give insight into perceived benefits, challenges and suggestions for improvement, allowing for improved therapeutic options for adolescents with anxiety. The feasibility method and outcomes will be guided by Orsmond and Cohn "The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions", and in line with the objectives, outcomes and interpretations of feasibility from Abbott and colleagues. Orsmond and Cohns highlights five objectives (A-E) that will be used as a template for assessing feasibility in our study. Our method for collecting data include questionnaires and user-data in the app from the patients, and qualitative interviews with both patients and clinicians. All outcomes will be reported in line with the CONSORT 2010 statement: extension to randomised pilot and feasibility trials, with adaptations to apply to our non-randomized feasibility trial.

2.1.1. Recruitment

The project aims to recruit 30 adolescents aged 13-18 from child and adolescent mental health services who, along with their clinicians, are willing to participate in the intervention as part of their treatment plan. All patient recruitment will be done in Helse Stavanger. The adolescents will receive gift cards of 250 NOK post assessment, and at 3-month follow-up. The adolescents that participate in qualitative interviews will receive an additional gift card of 250 NOK for their participation. Recruitment is set to begin in August 2025, with expected completion by the summer of 2026.

2.1.3 Procedures

Participants will first undergo a baseline assessment and be given guidance on how to use the Sidekick app to support anxiety exposure therapy. During the study period, all patients will be followed up through regular treatment at the Child and Adolescent Psychiatry Unit (BUP), which is usually weekly or bi-weekly. Patient responsibility and readiness will be maintained through this provider relationship as in regular treatment, but patients will also be provided with contact details for research personnel, who can then contact providers for the patients participating in the project. Exposure will mainly take place between treatment sessions, at times chosen by the youth themselves, or in collaboration with their clinician. Participants will undergo a baseline assessment online using the Youwell platform which is authorized for this purpose by Helse Vest. The assessment will be conducted at three timepoints: at baseline, at the end of treatment, and three months post-treatment. The feasibility and preliminary clinical outcomes of the intervention will be evaluated using quantitative methods before, during, and after the treatment. Additionally, qualitative interviews with therapists and patients will be conducted following the treatment to gather in-depth insights.

2.1.4 Interview guide

An interview guide will be used to gather data on participants' experiences, including perceived treatment. The interview guide will be developed in collaboration with users, and the interview is estimated to take 30 minutes to complete. Audio will be recorded using the app "Nettskjemadiktafon", which ensures safe storage of sensitive data. All data will be stored in TSD (in Norwegian, Service for Sensitive Data). The TSD service is designed for storing and post-processing sensitive data in compliance with the Norwegian "Personal Data Act" and "Health Research Act". Audio will be automatically transcribed using the service "Autotekst", and then manually checked by the PhD candidate.

2.1.5 Statistical analysis plan

As a feasibility study, no formal hypothesis testing will be conducted. Descriptive statistics will be used to summarize recruitment rates, retention rates, adherence, and data completeness to assess feasibility outcomes. Confidence intervals will be provided to estimate precision of feasibility parameters. Preliminary outcome measures will be explored to inform sample size calculations and study procedures for a future definitive trial. All analyses will be run using freely or commercially available software (R or SPSS statistics) by the applicant in collaboration with supervisors of the PhD-project. The sample size is based on recommendations for feasibility and pilot studies, recommending a sample size of 30 participants to establish feasibility.

2.1.6 Qualitative analysis plan

Using the NVivo software, qualitative data will be analyzed using thematic analysis to explore therapists' and users' experiences with the Sidekick app. Initial coding will capture key concepts, which will then be grouped into broader themes reflecting the core experiences of both therapists and adolescents. This process will highlight perceptions of the app, including its strengths and areas for improvement. Comparative analysis will contrast the themes from both perspectives to provide a comprehensive understanding of the app's impact and effectiveness in outpatient treatment. The findings will inform app enhancements and implementation strategies to better support therapists and adolescents in these settings.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 18 years old
* Adequate Norwegian reading, writing and speaking skills
* Access to the internett and a smart-phone
* Diagnosed anxiety disorder
* Receiving outpatient treatment for their anxiety disorder
* Exposure therapy included in therapy during the study period
* Therapist agrees to incorporate the app as an ad-on to therapy
* For patients receiving medication, inclusion requires a stable dose of medication for a psychiatric disorder for six weeks

Exclusion Criteria:

* Participants with serious mental illness, such as suicidality or poor general functioning may be excluded if participation is considered unfeasible or potentially harmful. Decision will be based on collaborative evaluation by the participants therapist and the research-team.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Sidekick app engagement and completion of tasks | From pre-treatment/baseline to post-treatment (variable and participant-dependent, estimated range: 4-12 weeks)
  Sidekick app engagement and completion of tasks will be evaluated through assessment of user-data from the app.
Credibility and Expectancy Questionnaire (CEQ-1) | At post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline)
  The Credibility and Expectancy Questionnaire (CEQ-1) is a 1-item self-report questionnaire used to assess treatment credibility and treatment expectancy.
  Minimum score: 1. Maximum score: 9. Higher scores mean better outcomes.
Client Satisfaction Questionnaire (CSQ-3) | At post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline)
  The Client Satisfaction Questionnaire (CSQ-3) is a 3-item self-report measure used clients satisfaction with a service. Minimum score: 1. Maximum score: 4. Higher scores mean better outcomes.
EuroQoL 5D-5L (EQ-5D-5L) | At pre-treatment/baseline and post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline)
  EuroQoL 5D-5L (EQ-5D-5L) is a self-report questionnaire assessing health-related quality of life and cost-effectiveness analysis. It assesses health on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Question 1-25: Minimum score: 1. Maximum score: 5. Higher scores mean worse outcomes. Question 26: Minimum score: 0. Maximum score: 100. Higher scores mean better outcomes.
Level of anxiety before, during and after exposure tasks | From pre-treatment/baseline to post-treatment (variable and participant-dependent, estimated range: 4-12 weeks) after every completed exposure task (variable and participant-dependent, estimated range: 1-20 exposure tasks per month)
  Participants will evaluate their level of anxiety on a sliding bar in the Sidekick app before, during and after every exposure task completed. User-data from the Sidekick app will be collected. Minimum score: 1. Maximum score: 10. Higher scores mean worse outcomes.
Recruitment | At pre-treatment/baseline.
  The investigators will assess recruitment capability and sample characteristics and provide a flow-chart to evaluate feasibility of completing the planned study.
Adherence | From pre-treatment/baseline to post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline), and from post-treatment to 3-month follow-up.
  The investigators will assess retention and follow-up rates, and adherence to procedures to evaluate feasibility of completing the planned study.
Qualitative interviews | At post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline).
  To evaluate user experiences from both patients and clinicians perspectives taking part in the study.
Revised Child Anxiety and Depression Scale (RCADS 47) | At pre-treatment/baseline, post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline), and 3-month follow-up.
  The Revised Child Anxiety and Depression Scale (RCADS) is a self-report measure of anxiety symptoms for children and adolescents aged 8-18 years old. It has 47 items, and results in subscales of separation anxiety, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder and major depressive disorder. The scale provides a total anxiety scale (sum of the 5 anxiety subscales) and a total internalizing scale (sum of all 6 subscales). Minimum score: 10 Maximum score: 3. Higher scores mean worse outcomes.
General self-efficacy scale (GSES) | At pre-treatment/baseline, post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline), and 3-month follow-up.
  The General self-efficacy scale (GSES) is a 10-item self-report questionnaire used to measure the respondents perceived self-efficacy. Minimum score: 1. Maximum score: 4. Higher scores mean better outcomes.
KIDSCREEN-10 | At pre-treatment/baseline, post-treatment (variable and participant-dependent, estimated range: 4-12 weeks post-baseline), and 3-month follow-up.
  KIDSCREEN-10 is a 10-item self-report questionnaire for children and adolescents aged 8-18 years old. It measures general health-related quality of life (HRQoL). Minimum score: 1. Maximum score: 5. Higher scores mean better outcomes.
Patient Exposure and Response Prevention Adherence Scale (PEAS) | From pre-treatment/baseline to post-treatment (variable and participant-dependent, estimated range: 4-12 weeks) after every completed exposure task (variable and participant-dependent, estimated range: 1-20 exposure tasks per month)
  The Patient Exposure and Response Prevention Adherence Scale (PEAS) is a 3-item self-report questionnaire designed to measure adherence of exposure and response prevention outside of therapy sessions. Minimum score: 0. Maximum score: 7. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander H Erga, PhD, Study Director — KORFOR, Helse Stavanger; Torgeir G Lid, PhD, Study Chair — KORFOR, Helse Stavanger; Emilie S Nordby, PhD, Study Chair — Forhelse, Helse Bergen; Tine Nordgreen, PhD, Study Chair — Forhelse, Helse Bergen; Pia R Hauge, Master, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger Universitetssykehus, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UngMeistring - About the project — https://forhelse.no/en/ungmeistring/about-the-project/